CLINICAL TRIAL: NCT01224626
Title: Zyvox (Linezolid) Special Investigation For Vancomycin-Resistant Enterococci (VRE)(Regulatory Post Marketing Commitment Plan)
Brief Title: Zyvox (Linezolid) Special Investigation For Vancomycin-Resistant Enterococci (VRE)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5951139
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-05

CONDITIONS: Vancomycin Resistance Enterococcus Faecium
Keywords: VRE; Japanese; Post Marketing Surveillance
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Zyvox (linezolid): Patients who have been treated with Zyvox (linezolid).
  Interventions: Drug: Zyvox (linezolid)

INTERVENTIONS:
Drug: Zyvox (linezolid) — Patients should be treated with Zyvox (linezolid) 600 mg every twelve hours.
  Other Names: linezolid, Zyvox

SUMMARY:
To collect the efficacy and safety information in subjects who have been treated with Zyvox (linezolid) for vancomycin resistance Enterococcus faecium infection for their appropriate use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject to whom Zyvox (linezolid) was administered.
* Infected subject with Vancomycin resistance Enterococcus faecium.

Exclusion Criteria:

* Infected subject with MRSA and other organism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who are prescribed to Zyvox (linezolid).
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951139&StudyName=Zyvox%20%28Linezolid%29%20Special%20Investigation%20For%20Vancomycin-Resistant%20Enterococci%20%28VRE%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional retrospective study.
Groups:
- Linezolid: Participants who have been treated with Zyvox (linezolid).
Period: Overall Study
Arm/Group | Linezolid
Started | 42
Completed | 41
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Linezolid
Number analyzed (Participants) | 41
Age, Customized [Number; unit: participants]
  <65 years | 12
  >=65 years | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 21
Past medical history [Number; unit: participants] — Past medical history is the patient's past experiences with illnesses, operations, injuries and treatments.
  The physician of this survey made the diagnosis or took from the participants.
  participants
    Present | 22
    Absent | 18
    Unknown | 1
Complications [Number; unit: participants] — Complications is the patient's current experiences with illnesses, operations, injuries and treatments.
  The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
  participants
    Present | 41
    Absent | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions.
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported as adverse events. Definition of adverse drug reaction was treatment related adverse events which were evaluated in company with the causal relationship to the investigational product.
Time Frame: Baseline to 8 weeks
Population: Safety analysis population consisted of the participants that satisfied the inclusion and exclusion conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 41
participants
  Platelet count decreased | 10
  Anaemia | 3
  White blood cell count decreased | 3
  Superinfection | 1
  Sepsis | 1
  Histiocytosis haematophagic | 1
  Pancytopenia | 1
  Dizziness postural | 1
  Neuropathy peripheral | 1
  Diarrhoea | 1
  Liver disorder | 1
  Renal disorder | 1
  Multi-organ failure | 1
  Aspartate aminotransferase increased | 1
  Haemoglobin decreased | 1
  Liver function test abnormal | 1
  Blood alkaline phosphatase increased | 1
  Red blood cell count decreased | 1

2. Secondary Outcome: Adverse Drug Reactions Unlisted in Japanese Package Insert.
Description: The adverse drug reactions that have not been included in Japanese package insert.
Time Frame: Baseline to 8 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 41
participants
  Sepsis | 1
  Histiocytosis haematophagic | 1
  Neuropathy peripheral | 1
  Liver disorder | 1
  Renal disorder | 1
  Multi-organ failure | 1

3. Primary Outcome: Number of Participants Categorized as Responders (Cure and Improved) to Zyvox (Linezolid) Treatment.
Description: Clinical overall effectiveness was evaluated by investigators based on clinical symptoms, laboratory test and investigator judgement, at the end of observation period. Clinical rating (cure/improved/not cured/unable to evaluate) was carried out. Definition of cured was disappearance of clinical symptom and/or Laboratory test abnormality. Definition of improved was improvement in clinical symptoms and/or laboratory test abnormality.
Time Frame: Baseline to 8 weeks
Population: The efficacy analysis population included all subjects from the safety analysis population in whom the efficacy of this drug could be evaluated.
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 17
participants | 16

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid
Serious Adverse Events (participants affected / at risk) | 9/41
Other Adverse Events (participants affected / at risk) | 21/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid (N=41)
Platelet count decreased (Investigations) | 5 (5)
White blood cell count decreased (Investigations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid (N=41)
Platelet count decreased (Investigations) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
White blood cell count decreased (Investigations) | 3 (3)
Superinfection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.